CLINICAL TRIAL: NCT01192347
Title: A Phase 4, Observational Study to Explore How Different Treatment Regimens Affect Continuation With Treatment in the First 6 Months Following Initiation of XAGRID Into Adult Patients' Essential Thrombocythemia Therapy
Brief Title: French Observational Xagrid (FOX) Study In Adult Patients With Essential Thrombocythemia
Acronym: FOX
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD422-702
Record Dates: First submitted 2010-08-26; First posted 2010-09-01 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Essential Thrombocythemia
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to explore how different treatment regimens affect continuation with treatment in the first 6 months following initiation of XAGRID into adult patients' essential thrombocythemia therapy.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 18 years and older.
2. High-risk ET Patients, uncontrolled by first-line (or previous) cytoreductive treatment for efficacy or tolerance reasons.
3. Patients who have been on second- or third-line XAGRID treatment for up to 1 month, or for whom a decision has been documented to commence second line XAGRID treatment.
4. Patients able to understand and able and willing to participate in the study, and provide a personally dated and signed written informed consent form.

Exclusion Criteria

1. Patients with a known or suspected intolerance or hypersensitivity to XAGRID, closely related compounds, or any of the stated ingredients.
2. Patients for whom there is an intention to treat with combinations of cytoreductive therapy.
3. Patients participating in a separate clinical trial where their treatment is defined by that study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2012-12-21 (Actual); Study Completion 2012-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- France (46):
  - GH Pitie Salpetriere, Paris, Cedex 13
  - CH DU Pays D Aix, Aix-en-Provence, Cedex 1
  - Hopital Dupuytren, Limoges, Cedex 1
  - Hopital Emile Muller, Mulhouse, Cedex 1
  - Hopital Hotel Dieu Et Hme, Nantes, Cedex 1
  - Hopital Tenon, Paris, Cedex 20
  - Nouvelles Cliniques Nantaises, Nantes, Cedex 2
  - Hopital Hautepierre, Strasbourg, Cedex 2
  - Hopital De L Archet, Nice, Cedex 3
  - Clinique Du Parc, Caen, Cedex 4
  - Hotel Dieu, Angers, Cedex 9
  - CH Departemental Des Oudairies, La Roche-sur-Yon, Cedex 9
  - Hopital Pontchaillou, Rennes, Cedex 9
  - Hia Sainte Anne, Toulon, Cedex 9
  - Ch D Arras, Arras, Cedex
  - Hopital Robert Ballanger, Aulnay-sous-Bois, Cedex
  - CH De Blois, Blois, Cedex
  - Ch De Fleyriat, Bourg-en-Bresse, Cedex
  - CME, Brest, Cedex
  - Hopital Augustin Morvan, Brest, Cedex
  - Ch De Brive La Gaillarde, Brive-la-Gaillarde, Cedex
  - Hopital Henri Mondor, Créteil, Cedex
  - CH De Bicetre, Le Kremlin-Bicêtre, Cedex
  - CHRU Lille - Hopital Huriez, Lille, Cedex
  - Hopital Saint Philibert, Lomme, Cedex
  - Hopital Edouard Herriot, Lyon, Cedex
  - Institut J Paoli Calmettes, Marseille, Cedex
  - Hopital N D Bon Secours, Metz, Cedex
  - Clinique Pont de Chaume, Montauban, Cedex
  - Hopital Saint Antoine, Paris, Cedex
  - GH Pitie Salpetriere, Paris, Cedex
  - Hopital Saint Jean, Perpignan, Cedex
  - Hopital De Haut Leveque, Pessac, Cedex
  - CHI Poissy Saint German en Laye, Poissy, Cedex
  - Chi De Cornouaille, Quimper, Cedex
  - Hopital de La Maison Blanche, Reims, Cedex
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez, Cedex
  - Hopital Font Pre, Toulon, Cedex
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy, Cedex
  - Ch De Vendome, Vendôme, Cedex
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Robert Boulin, Libourne
  - CHU Nord - Chemin Des Bourrely, Marseille
  - CHRA, Metz-Tessy
  - Cabinet D'Hematologie, Perpignan
  - Centre De Radiotherapie, Strasbourg

REFERENCES:
- [Derived] Rey J, Viallard JF, Keddad K, Smith J, Wilde P, Kiladjian JJ; FOX study investigators. Characterization of different regimens for initiating anagrelide in patients with essential thrombocythemia who are intolerant or refractory to their current cytoreductive therapy: results from the multicenter FOX study of 177 patients in France. Eur J Haematol. 2014 Feb;92(2):127-36. doi: 10.1111/ejh.12210. Epub 2013 Nov 25. PMID 24118452

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 177 subjects were enrolled, but 2 never received Anagrelide Hydrochloride (Xagrid) and were excluded from the trial (n = 175).
Groups:
- Anagrelide Hydrochloride: The decision to initiate Anagrelide Hydrochloride and the dose prescribed was made by treating physician.
Period: Overall Study
Arm/Group | Anagrelide Hydrochloride
Started | 175
Completed | 163
Not Completed | 12
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Suspected serious adverse drug reaction | 1
Not completed — Patient seen in different hospital | 1
Not completed — Patient not visiting hospital regularly | 1
Not completed — Patient did not show up for visits | 1

BASELINE CHARACTERISTICS:
Population: Safety Set was used for Baseline measures. Safety Set comprised all patients who had taken at least 1 dose of Anagrelide Hydrochloride and had at least 1 post-baseline safety assessment. Two patients did not receive Anagrelide Hydrochloride, therefore n = 175 for the Safety Set.
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (15.4)
Age, Customized [Count of Participants; unit: Participants]
  <=60 years | 42
  >60 years | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 67
Region of Enrollment [Count of Participants; unit: Participants] — Enrolled participants who received at least 1 dose of XAGRID
  Participants
    France | 175

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Continuation of Anagrelide Hydrochloride at 6 Months: Withdrawal of Previous Cytoreductive Therapy Before Anagrelide Hydrochloride Initiation
Description: Patients who had taken a previous cytoreductive therapy were divided into subgroups based on the treatment regimens used when Anagrelide Hydrochloride treatment was initiated, using the following variables: •Withdrawal of previous cytoreductive therapy: -Before: if a stop date of previous cytoreductive therapy was prior to the date of Anagrelide Hydrochloride initiation -After: if a stop date of previous cytoreductive therapy was between the first administration and the last administration of Anagrelide Hydrochloride during the follow-up -Not Withdrawn: in all other cases
Time Frame: 6 months
Population: Full Analysis Set (FAS) comprised all enrolled patients for whom Anagrelide Hydrochloride therapy was initiated. Subjects who had not taken any previous cytoreductive therapy other than Anagrelide Hydrochloride were excluded from the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 115
percentage of subjects | 81.7 [73.5 to 88.3]

2. Primary Outcome: Percentage of Subjects With Continuation of Anagrelide Hydrochloride at 6 Months: Withdrawal of Previous Cytoreductive Therapy After Anagrelide Hydrochloride Initiation
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 39
percentage of subjects | 94.9 [82.7 to 99.4]

3. Secondary Outcome: Percentage of Subjects With Anagrelide Hydrochloride Starting Doses
Time Frame: 6 months
Population: Safety Set comprised all subjects who had taken at least 1 dose of Anagrelide Hydrochloride and had at least 1 post-baseline safety assessment documented.
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 175
percentage of subjects
  0.3 mg/day | 0.6
  0.5 mg/day | 41.1
  1.0 mg/day | 52.6
  1.3 mg/day | 0.6
  1.5 mg/day | 5.1

4. Secondary Outcome: Number of Subjects With Anagrelide Hydrochloride Titration Modifcations- First Modification Only
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 175
participants
  -1.0 mg/day | 1
  -0.5 mg/day | 7
  -0.2 mg/day | 2
  No change | 26
  +0.2 mg/day | 1
  +0.5 mg/day | 109
  +1.0 mg/day | 12
  +1.2 mg/day | 1
  Dose interruption | 9
  Discontinued therapy | 7

5. Primary Outcome: Percentage of Subjects With Continuation of Anagrelide Hydrochloride at 6 Months: No Withdrawal of Previous Cytoreductive Therapy
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 16
percentage of subjects | 81.3 [54.4 to 96.0]

6. Primary Outcome: Percentage of Subjects With Continuation of Anagrelide Hydrochloride at 6 Months: When the Dosing Was Consistent With the Summary of Product Characteristics (SmPC)
Description: Patients who had taken a previous cytoreductive therapy were divided into subgroups based on the treatment regimens used when XAGRID treatment was initiated, using the following variables: •Initiation of XAGRID dosing consistent with the Summary of Product Characteristics (SmPC): •Consistent if: -The starting dose was <=1 mg/day, AND -Any increase in dose was no more than 0.5mg/day, AND -Any increase in dose was made at least 7 days after first initiation or at least 7 days after any previous modification (up or down), AND -The maximum dose did not exceed 10 mg/day at any stage. •Inconsistent: in all other cases
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 133
percentage of subjects | 83.5 [76.0 to 89.3]

7. Primary Outcome: Percentage of Subjects With Continuation of Anagrelide Hydrochloride at 6 Months: When the Dosing Was Inconsistent With the Summary of Product Characteristics (SmPC)
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 37
percentage of subjects | 89.2 [74.6 to 97.0]

8. Primary Outcome: Percentage of Subjects Achieving Platelet Target Response: Withdrawal of Previous Cytoreductive Therapy Before Anagrelide Hydrochloride Initiation
Description: Full response is a platelet count of <400x10^9/L. Partial response is a platelet count between 400-600x10^9/L or a platelet count reduction of 200x10^9. Patients who had taken a previous cytoreductive therapy were divided into subgroups based on the treatment regimens used when Anagrelide Hydrochloride treatment was initiated, using the following variables: •Withdrawal of previous cytoreductive therapy: -Before: if a stop date of previous cytoreductive therapy was prior to the date of Anagrelide Hydrochloride initiation -After: if a stop date of previous cytoreductive therapy was between the first administration and the last administration of Anagrelide Hydrochloride during the follow-up -Not Withdrawn: in all other cases
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 115
percentage of subjects
  Full response | 41.7 [32.6 to 51.3]
  Partial response | 25.2 [17.6 to 34.2]

9. Primary Outcome: Percentage of Subjects Achieving Platelet Target Response: Withdrawal of Previous Cytoreductive Therapy After Anagrelide Hydrochloride Initiation
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 39
percentage of subjects
  Full response | 48.7 [32.4 to 65.2]
  Partial response | 38.5 [23.4 to 55.4]

10. Primary Outcome: Percentage of Subjects Achieving Platelet Target Response: No Withdrawal of Previous Cytoreductive Therapy
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 16
percentage of subjects
  Full response | 25.0 [7.3 to 52.4]
  Partial response | 31.3 [11.0 to 58.7]

11. Primary Outcome: Percentage of Subjects Achieving Platelet Target Response: When the Dosing Was Consistent With the Summary of Product Characteristics (SmPC)
Description: Full response is a platelet count of <400x10^9/L. Partial response is a platelet count between 400-600x10^9/L or a platelet count reduction of 200x10^9. Patients who had taken a previous cytoreductive therapy were divided into subgroups based on the treatment regimens used when XAGRID treatment was initiated, using the following variables: •Initiation of XAGRID dosing consistent with the Summary of Product Characteristics (SmPC): •Consistent if: -The starting dose was <=1 mg/day, AND -Any increase in dose was no more than 0.5mg/day, AND -Any increase in dose was made at least 7 days after first initiation or at least 7 days after any previous modification (up or down), AND -The maximum dose did not exceed 10 mg/day at any stage. •Inconsistent: in all other cases
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 133
percentage of subjects
  Full response | 44.4 [35.8 to 53.2]
  Partial response | 30.8 [23.1 to 39.4]

12. Primary Outcome: Percentage of Subjects Achieving Platelet Target Response: When the Dosing Was Inconsistent With the Summary of Product Characteristics (SmPC)
Description: as for outcome 11
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 37
percentage of subjects
  Full response | 32.4 [18.0 to 49.8]
  Partial response | 21.6 [9.8 to 38.2]

13. Secondary Outcome: Summary of Adverse Drug Reactions (ADR): Withdrawal of Previous Cytoreductive Therapy Before Anagrelide Hydrochloride Initiation
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 115
percentage of subjects
  ADR | 44.3
  Serious ADR | 5.2
  ADR leading to stopping Xagrid | 16.5

14. Secondary Outcome: Summary of Adverse Drug Reactions: Withdrawal of Previous Cytoreductive Therapy After Anagrelide Hydrochloride Initiation
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 39
percentage of subjects
  ADR | 51.3
  Serious ADR | 2.6
  ADR leading to stopping Xagrid | 15.4

15. Secondary Outcome: Summary of Adverse Drug Reactions: No Withdrawal of Previous Cytoreductive Therapy
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 16
percentage of subjects
  ADR | 37.5
  Serious ADR | 6.3
  ADR leading to stopping Xagrid | 12.5

16. Secondary Outcome: Summary of Adverse Drug Reactions: When the Dosing Was Consistent With the Summary of Product Characteristics (SmPC)
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 133
percentage of subjects
  ADR | 39.1
  Serious ADR | 4.5
  ADR leading to stopping Xagrid | 18.8

17. Secondary Outcome: Summary of Adverse Drug Reactions: When the Dosing Was Inconsistent With the Summary of Product Characteristics (SmPC)
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 37
percentage of subjects
  ADR | 67.6
  Serious ADR | 5.4
  ADR leading to stopping Xagrid | 5.4

18. Secondary Outcome: Maximum Daily Dose of Anagrelide Hydrochloride
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 175
mg/day | 1.5 (0.6)

ADVERSE EVENTS:
Arm/Group | Anagrelide Hydrochloride
Serious Adverse Events (participants affected / at risk) | 8/175
Other Adverse Events (participants affected / at risk) | 81/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide Hydrochloride (N=175)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anagrelide Hydrochloride (N=175)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Edema peripheral (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 22 (24)
Tachycardia (Cardiac disorders) | 5 (5)
Tinnitis (Ear and labyrinth disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 10 (10)
Headache (Nervous system disorders) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.